CLINICAL TRIAL: NCT04963985
Title: The Effect of Tafamidis on Transthyretin Stabilization, Safety, Tolerability and Efficacy in Transthyretin Amyloid Polyneuropathy Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2020466
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related | interventions — tafamidis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafamidis group (Experimental): During the treatment period, each participant will receive 20 mg tafamidis meglumine once daily for 24 weeks.
  Interventions: Drug: Tafamidis Pill

INTERVENTIONS:
Drug: Tafamidis Pill — Oral

SUMMARY:
Transthyretin amyloid polyneuropathy (ATTR-PN) is a fatal illness resulting from autosomal dominantly inherited single-point mutations on the transthyretin gene.

Tafamidis is a specific stabilizer of both variant and wild-type TTR. Tafamidis binds to TTR at the thyroxine binding sites and inhibits TTR tetramer dissociation, the rate limiting step in the amyloidogenic process. The result disrupts the amyloid cascade and fibril formation and interrupts disease progression.

This study provides the basis for the study of the effect of tafamidis on the stability of transthyretin and its safety, tolerance and efficacy in patients with transthyretin amyloid polyneuropathy.

DETAILED DESCRIPTION:
Transthyretin amyloidosis is a protein misfolding disease with a broad spectrum of manifestations. When the peripheral nerves are affected predominately, the disease is termed transthyretin amyloid polyneuropathy (ATTR-PN). When the heart is primarily affected, the disease is called transthyretin amyloid cardiomyopathy (ATTR-CM). ATTR-PN is a fatal illness resulting from autosomal dominantly inherited single-point mutations on the transthyretin gene.

Tafamidis is a specific stabilizer of both variant and wild-type TTR. Tafamidis binds to TTR at the thyroxine binding sites and inhibits TTR tetramer dissociation, the rate limiting step in the amyloidogenic process. The result disrupts the amyloid cascade and fibril formation and interrupts disease progression.

In China, ATTR-PN is rare, estimated at approximately 1997 persons . In recent years, about 30-40 case reports have been published and several ATTR-PN families were reported with different TTR gene mutations from those observed in Europe. Delay in the time to diagnosis is a major obstacle to the optimal management of ATTR-PN in China, and patients will typically wait several years between the emergence of first clinical signs and receiving an accurate diagnosis. There is a critical need to raise disease awareness, to facilitate earlier diagnosis and an urgency to enable access to treatment given the significant unmet medical need in this rare and fatal disease.

ELIGIBILITY:
Inclusion Criteria:

-

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Male or female participants between the ages of 18 and 80 years.

   Type of Participant and Disease Characteristics:
2. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures.
3. Participants have amyloid documented by biopsy in accordance with institutional site standard of care (Biopsy must have been performed within 5 years of enrollment).
4. Participants must have a TTR mutation that is associated with ATTR-PN. (See Section 8.2.6.3 for further details).
5. Participants have peripheral and/or autonomic neuropathy with a Karnofsky Performance Status ≥50 (refer to Appendix 5).
6. Stages of disease according to symptom severity-stage I.

   Informed Consent:
7. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

-

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions:

1. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

   Prior/Concomitant Therapy:
2. Chronic use of non-protocol approved non-steroidal anti-inflammatory drugs (NSAIDs), defined as greater than 3-4 times/month. The following NSAID are allowed: acetylsalicylic acid, etodolac, ibuprofen, indomethacin, ketoprofen, nabumetone, naproxen, nimesulide, piroxicam, and sulindac.
3. Use of diflunisal, tauroursodeoxycholate, doxycycline or a TTR stabilizing agent, or other experimental interventions for familial amyloidosis within 30 days prior to the study entry and/or during study participation. Participants who are taking or who have previously taken tafamidis.
4. Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).

   Diagnostic Assessments:
5. Participant has primary (light chain) or secondary amyloidosis.
6. If female, participant is pregnant or breast feeding, or plans to be pregnant or breast feeding in the next 18 months.
7. Participant has received prior liver or any other organ except cornea transplantation.
8. Participant has no recordable sensory threshold for vibration perception in both feet, as measured by CASE IV or participant requires significant assistance with ambulation or is wheel chair bound.
9. Participants with positive results for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), and/or human immunodeficiency virus (HIV).
10. Participant has liver function test abnormalities: alanine transaminases (ALT) and/or aspartate transaminases (AST) >2 times upper limit of normal (ULN) that in the medical judgment of the investigator are due to reduced liver function or active liver disease.
11. Participants with cardiomyopathy specific TTR mutations (Val122Ile, Leu111Met, Ile68Leu).
12. Participant has a co-morbidity anticipated to limit survival to less than 18 months.
13. Participant has other causes of sensorimotor neuropathy (B12 deficiency, Diabetes Mellitus, HIV treated with retroviral medications, thyroid disorders, alcohol abuse, Fabry disease, Lyme disease, sarcoidosis, Sjogren's Syndrome, Systemic Lupus Erythematosus, alcohol dependency, celiac disease, Chronic Inflammatory Demyelinating Polyneuropathy, and chronic inflammatory diseases).

    Other Exclusions:
14. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
TTR stabilization compared with Baseline | at Week 8
  TTR stabilization at Week 8 compared with Baseline, as measured by a validated immunoturbidimetric assay.

SECONDARY OUTCOMES:
TTR stabilization | each follow up visit after Week 8（Week 8, Week 12 and Week 24）
  TTR stabilization at Week 8 compared with Baseline, as measured by a validated immunoturbidimetric assay.
TTR concentration | at Day 1(baseline), Week 8, Week 12 and Week 24
Neuropathy Impairment Score：NIS-LL (lower limb) | at Day 1(baseline) and Week 24
  Change from baseline
TQOL score and 5 domains as measured by the Norfolk QOL - Diabetic Neuropathy (Norfolk QOL-DN) | at Day 1(baseline) and Week 24
  Change from baseline
TQOL score and 5 domains asmeasured by the Norfolk | at Day 1(baseline) and Week 24
  Change from baseline
"Σ7 NTs NDS" as measured by nerve conduction studies (NCS), vibration detection threshold (VDT) and heart rate response to deep breathing (HRDB). | at Day 1(baseline) and Week 24
  Change from baseline
Modified Body Mass Index (mBMI). | at Day 1(baseline) and Week 24
  Change from baseline
36-item survey form (SF-36). | at Day 1(baseline) and Week 24
  Change from baseline
EQ-5D-5L Index Score. | at Day 1(baseline) and Week 24
  Change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No